CLINICAL TRIAL: NCT02096289
Title: A Phase I Trial Evaluating Oral Thioridazine in Combination With Intermediate Dose Cytarabine in Patients 55 Years and Older With Acute Myeloid Leukemia Who Have Relapsed or Have Refractory Disease
Brief Title: Safety Study of Thioridazine in Combination With Cytarabine to Treat Relapsed or Refractory Acute Myeloid Leukemia
Acronym: THORIDAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Juravinski Cancer Centre Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2013-THORIDAL
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Thioridazine; Phase I; Clinical Trial
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Thioridazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thioridazine (Experimental): Up to 3 dose levels of thioridazine will be assessed sequentially: 25 mg Q6H (Level I), 50 mg Q6H (Level II) and 100 mg Q6H (Level III). The duration of thioridazine therapy is for a total of 21 days (Days 1-22 on study). All patients will receive cytarabine 1 g/m2 administered as a 2 hour infusion for 5 consecutive days (Days 6-10 on study).
  Interventions: Drug: Thioridazine

INTERVENTIONS:
Drug: Thioridazine

SUMMARY:
This is a Phase I trial investigating the safety of using thioridazine in addition to cytarabine in elderly patients with relapsed or refractory Acute Myeloid Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of AML according to the WHO Classification1
* AML is refractory or relapsed (requiring at least 5% leukemic blasts in the bone marrow, regardless of the presence of other features such as new or recurrent dysplastic changes or extra medullary disease) according to the following definitions:

  * Relapsed (defined as ≥ 5% leukemic blasts in the bone marrow) after three months from receiving up to three prior induction regimens.
  * Refractory (defined as ≥ 5% leukemic blasts in the bone marrow) to not more than one prior induction regimen (defined as failure to achieve a CR or CRi following induction therapy).
* 55 years of age or older.

Exclusion Criteria:

* Receiving any other systemic anti-leukemic therapy (standard or investigational).
* Having received more than two prior chemotherapy lines for AML. Induction/consolidation therapy and bone marrow transplant are each considered a line of therapy.
* Having received previous AML therapy within four weeks of the first dose of study drug, with the exception of hydroxyurea.
* Clinical evidence suggestive of CNS involvement with leukemia unless a lumbar puncture confirms the absence of leukemic blasts in the CSF.
* Acute promyelocytic leukemia.
* An ECOG performance status of 3 or more.
* Inadequate renal function (i.e., estimated GFR < 60 mL/min/1.73m2).
* Inadequate hepatic function (i.e., serum bilirubin > 1.5×ULN; AST, ALT and alkaline phosphatase > 2.5×ULN).
* Presence of acute or chronic GVHD.
* Presence of a systemic fungal, bacterial, viral or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Having any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo induction therapy.
* Diagnosed with a condition that can prolong the QT interval (e.g., long QT syndrome) or have a QTc interval ≥ 470ms if male, or ≥ 480ms if female.
* Left ventricular ejection fraction less than 45%.
* History of uncontrolled cardiac arrhythmia.
* Known severe hypotensive or hypertensive heart disease.
* Prior malignancy, unless the patient has been disease-free for at least five years following curative intent therapy, with the following exceptions: Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, if definitive treatment for the condition has been completed; or patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values if hormonal therapy has been initiated or a radical prostatectomy has been performed.
* Known HIV positivity.
* Known pregnancy or lactating female.
* Presence of a psychiatric disorder that would interfere with consent, study participation, or follow-up.
* Unable to provide informed consent.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 36 days
  Both acute and late toxicities will be determined according to NCI-CTCAE version 4.03

SECONDARY OUTCOMES:
Assessment of Functional Leukemia Stem Cells | Up to 36 days
  Bone marrow and peripheral blood samples obtained from patients treated with thioridazine and cytarabine will be analyzed in four separate assays.
Pharmacokinetic Analysis of Thioridazine Serum Trough Levels | Up to 36 days
  Pharmacokinetic modeling will be performed to estimate values for individual C min levels.
Assessment of Objective Tumor Response | Up to 36 days
  Tumor responses are categorized as either a complete remission, a complete remission with incomplete count recovery, a partial remission, a treatment failure, or as not evaluable
Pharmacogenetic Analysis of Thioridazine Serum Trough Levels | Up to 36 days
  Cytochrome P450 2D6 genotype will be determined to examine genetic contribution to thioridazine Cmin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mark N Levine, MD, Study Director — Ontario Clinical Oncology Group, McMaster University; Ronan Foley, MD, Principal Investigator — Hamilton Health Sciences, McMaster University
Locations (1):
- Juravinski Hospital & Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Aslostovar L, Boyd AL, Almakadi M, Collins TJ, Leong DP, Tirona RG, Kim RB, Julian JA, Xenocostas A, Leber B, Levine MN, Foley R, Bhatia M. A phase 1 trial evaluating thioridazine in combination with cytarabine in patients with acute myeloid leukemia. Blood Adv. 2018 Aug 14;2(15):1935-1945. doi: 10.1182/bloodadvances.2018015677. PMID 30093531